CLINICAL TRIAL: NCT04316780
Title: Impact of Pre-transplant Anti-fibrotic Therapy for Idiopathic Pulmonary Fibrosis Upon Lung Transplant Outcomes
Brief Title: Impact of Pre-transplant Anti-fibrotic Therapy for IPF Upon Lung Transplant Outcomes
Acronym: IPF-LTOS
Status: Completed | Type: Observational
Sponsor: Steward St. Elizabeth's Medical Center of Boston, Inc. (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Peter LaCamera, Chief of Pulmonary, Critical Care and Sleep Medicine, Steward St. Elizabeth's Medical Center of Boston, Inc.
Other Study IDs: IPF-LTOS
Record Dates: First submitted 2019-04-18; First posted 2020-03-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Lung Transplant; Nintedanib; Pirfenidone; IPF
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Nintedanib until 0 day - 2 days before transplant: Nintedanib taken until 0 - 2 days before receiving transplant
  Interventions: Other: Retrospective observational study- no intervention to occur.
- Nintedanib until 3 days - 28 days before transplant: Nintedanib taken until 3-28 days before receiving transplant
  Interventions: Other: Retrospective observational study- no intervention to occur.
- Nintedanib until > 28 days before transplant: Nintedanib taken until more than 28 days before receiving transplant
  Interventions: Other: Retrospective observational study- no intervention to occur.
- Pirfenidone until 0 day - 1 day before transplant: Pirfenidone taken until 0 - 1 day before receiving transplant
  Interventions: Other: Retrospective observational study- no intervention to occur.
- Pirfenidone until 2 days - 28 days before transplant: Pirfenidone taken until 2-28 day before receiving transplant
  Interventions: Other: Retrospective observational study- no intervention to occur.
- Pirfenidone until > 28 days before transplant: Pirfenidone taken more than 28 days before receiving transplant
  Interventions: Other: Retrospective observational study- no intervention to occur.

INTERVENTIONS:
Other: Retrospective observational study- no intervention to occur. — Subject data will be grouped based on the anti-fibrotic medication at the time of lung transplant listing eligibility and when medication was stopped relative to the transplant.

SUMMARY:
Two oral medications, nintedanib and pirfenidone, were approved simultaneously by the FDA in October 2014 for the treatment of this disease. They are both considered anti-fibrotic agents and they each proved to slow the progression of disease in their respective clinical trials. Because of their anti-fibrotic properties, there have been concerns about the potential of these medications to impair wound healing following surgery. These concerns have led to variable approaches with respect to the management of the medications in patients listed for lung transplantation.

It is unknown whether continuing anti-fibrotic medications until the time of transplant increases the risks of intra-operative and post-transplant complications. Conversely, there are concerns that stopping the medications prematurely may promote a more rapid clinical decline in those awaiting transplantation and increase risk of death while on waiting lists. Whether there is a risk or benefit of continuing the medications during the pre-transplant period deserves investigation with the goal of establishing guidelines and best-practices. Once more is known about how best to manage anti-fibrotic therapy in the pre-transplant period, the question of whether these medications should be restarted following transplantation will also ultimately deserve exploration.

DETAILED DESCRIPTION:
Idiopathic pulmonary fibrosis (IPF) is a terminal illness that typically develops in the sixth and seventh decades of life. It is a relentless fibrotic parenchymal lung disease that results in restrictive physiology and worsening symptoms of cough and shortness of breath. The median life expectancy from the time of diagnosis is in the 3-5 year range. The only therapy that has proven to extend life expectancy is lung transplantation.

There are 3 relevant, unanswered questions pertaining to the use of anti-fibrotic therapy for IPF around the time of lung transplantation:

1. Does stopping the medications prematurely while awaiting lung transplantation result in a greater risk of death due to acceleration of IPF?
2. Does continuing the medications until the time of transplant increase the risk of intra- and/or post-operative complications?
3. Is there a role for post-transplant anti-fibrotic therapy to reduce complications such as stenosis of the anastomosis, bronchiolitis obliterans syndrome and restrictive allograft syndrome, and/or to preserve native lung function following a single lung transplant?

The primary goal of this observational, pilot study is to collect retrospective data with the intention of using the findings to select primary outcomes and determine sample size for a sufficiently powered subsequent study.

The investigators will focus on the following aims:

Aim 1: Assess whether the time period between discontinuation of anti-fibrotic therapy for IPF and lung transplantation impacts (a) the risk of intra-operative and post-transplant complications and (b) short term survival.

Aim 2: Explore whether discontinuing anti-fibrotic therapy prior to lung transplantation is associated with increased risk of death while awaiting a transplant.

At the participating sites, all patients with IPF listed for lung transplantation who were being treated with one of the 2 anti-fibrotic therapies continuously for at least 90 days at the time of their eligibility for listing will be included. Outcomes include events that occurred after being listed and while waiting for lung transplantation, intra-operative and peri-operative events, and mortality data out to 6 months. Patients that underwent additional interventions (coronary artery bypass grafting, valve replacement) at the time of their transplant will be excluded.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of IPF
2. Taking one of the two anti-fibrotic therapies (nintedanib or pirfenidone) continuously for at least 90 days at the time of eligibility for listing
3. Listed for lung transplantation between July 1, 2015 and June 30, 2019

Exclusion Criteria:

1. Patients that underwent additional interventions (i.e. coronary artery bypass grafting, valve replacement) at the time of their lung transplant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with IPF listed for lung transplantation who were being treated with one of the 2 anti-fibrotic therapies continuously for at least 90 days at the time of their eligibility for listing will be included.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Lung transplant complications | 6 months
  The proportions of patients in each group who develop (a) intra-operative outcomes and complications (need for ECMO/cardiopulmonary bypass and blood transfusions) and (b) post-transplant outcomes and complications (mechanical ventilation days, number of days with air leak and chest tube, primary graft dysfunction, anastomotic dehiscence, wound dehiscence, sternal breakdown / dehiscence, post-op infection, post-operative return to OR, blood transfusions) will be calculated.
Short term survival | 6 months
  Post-transplant, patients will be followed for six months to estimate the mean, median, and variability of short-term survival in each group.
Patient deaths while awaiting a transplant | From date of listed for transplant until the date of death from any cause assessed up to 54 months.
  The proportion of patients in each of the six groups who die after being listed and prior to receiving a transplant.
Disease progression while awaiting a transplant | From date of listed for transplant until the date of transplant or date of death from any cause assessed up to 54 months.
  Changes in forced vital capacity (FVC) as measured in liters will be compared between groups.
Disease progression while awaiting a transplant | From date of listed for transplant until the date of transplant or date of death from any cause assessed up to 54 months.
  Changes in percent predicted forced vital capacity (FVC%) as measured in percentage will be compared between groups.
Disease progression while awaiting a transplant | From date of listed for transplant until the date of transplant or date of death from any cause assessed up to 54 months.
  Changes in diffusing capacity of the lung for carbon monoxide (DLCO) as measured in ml/mmHg/min will be compared between groups.
Disease progression while awaiting a transplant | From date of listed for transplant until the date of transplant or date of death from any cause assessed up to 54 months.
  Changes in percent predicted diffusing capacity of the lung for carbon monoxide (DLCO%) as measured in percentage will be compared between groups.
Disease progression while awaiting a transplant | From date of listed for transplant until the date of transplant or date of death from any cause assessed up to 54 months.
  Changes in Lung Allocation Score (scale from 0-100; higher score reflecting higher priority for transplant) will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Peter LaCamera, M.D., Principal Investigator — St. Elizabeth's Medical Center
Locations (8):
- United States (8):
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Astor TL, Goldberg HJ, Snyder LD, Courtwright A, Hachem R, Pena T, Zaffiri L, Criner GJ, Budev MM, Thaniyavarn T, Leonard TB, Bender S, Barakat A, Breeze JL, LaCamera P. Anti-fibrotic therapy and lung transplant outcomes in patients with idiopathic pulmonary fibrosis. Ther Adv Respir Dis. 2023 Jan-Dec;17:17534666231165912. doi: 10.1177/17534666231165912. PMID 37073794